CLINICAL TRIAL: NCT06200129
Title: İmportance of Scattered White Spots Detected in the Duodenum and Their Relationship wıth Zonulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Semih Sezer, clinic physician, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: zonulinsws
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Duodenal Diseases; White Spot Lesion
MeSH Terms: conditions — Duodenal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sws grade 1 (Experimental): The group that defined as scattered white spots on the normal duodenal mucosa that could not be wiped away by washing, appearing as white spots
  Interventions: Diagnostic Test: sws grade 1
- sws grade 2 (Experimental): The group that defined as a diffuse or patchy white appearance on villi that could not be wiped away by washing on the mucosa.
  Interventions: Diagnostic Test: sws grade 2
- control (Experimental): The group with a normal appearance of the duodenal mucosa, where scattered white spots were not detected.
  Interventions: Diagnostic Test: control

INTERVENTIONS:
Diagnostic Test: sws grade 1 — Blood for zonulin level was drawn from the group of patients with typical white lesions in the duodenum, called grade 1.
  Arms: sws grade 1
Diagnostic Test: sws grade 2 — Blood for zonulin level was drawn from the group of patients with typical white lesions in the duodenum, called grade 2
  Arms: sws grade 2
Diagnostic Test: control — Group of patients without scattered white lesions in the dueodenum on endoscopy.
  Arms: control

SUMMARY:
With our study, we aimed to determine whether there is a correlation between zonulin, which plays a crucial role in intestinal barrier function and is implicated in the etiopathogenesis of many chronic and autoimmune diseases, and scattered white spots lesions associated with lymphatic stasis and inflammation in the duodenum.

DETAILED DESCRIPTION:
During esophagogastroduodenoscopy (EGD), rarely encountered lesions in the duodenum present as scattered white spots (SWS) on the normal mucosa. Although not fully understood in terms of specific association with any particular disease and clinical significance, some studies have often observed chronic non-specific duodenitis (CND) and intestinal lymphangiectasia (IL) in lesions with SWS. This condition is thought to be related to lymphatic stasis.

Patients included 63 individuals with identified SWS during EGD and 30 patients with a normal appearance of the duodenal mucosa were selected as the control group. SWS lesions were categorized into two groups, grade 1 and grade 2, based on the degree of density and endoscopic appearance. Biopsies were taken from the duodenum, antrum, and corpus. It was examined for IL, CND, giardiasis, and villous atrophy. Venous blood samples were collected from all patients for serum zonulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scattered white patchy lesions in the duodenum on endoscopy and control group patients with normal duodenum on endoscopy.

Exclusion Criteria:

* active gastroenteritis
* acute kidney failure
* chronic kidney failure
* type-1 diabetes
* inflammatory bowel disease
* duodenal ulcer,
* duodenal tumor
* autoimmune diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
zonulin levels | immediately after the procedure
  Patients with scattered white spots in the duodenum had blood drawn for zonulin level immediately after the procedure.

SECONDARY OUTCOMES:
Duodenal and gastric pathologic conditions | During the endoscopy
  Biopsies from the duodenum and gastric antrum and corpus were taken during the endoscopy from patients with scattered white spots in the duodenum.

CONTACTS AND LOCATIONS:
Overall Officials: semih sezer, Principal Investigator — clinic physician
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tas A, Koklu S, Beyazit Y, Akbal E, Kocak E, Celik H, Biyikoglu I. The endoscopic course of scattered white spots in the descending duodenum: a prospective study. Gastroenterol Hepatol. 2012 Feb;35(2):57-64. doi: 10.1016/j.gastrohep.2011.11.010. Epub 2012 Jan 20. PMID 22260755
- [Result] Fasano A, Shea-Donohue T. Mechanisms of disease: the role of intestinal barrier function in the pathogenesis of gastrointestinal autoimmune diseases. Nat Clin Pract Gastroenterol Hepatol. 2005 Sep;2(9):416-22. doi: 10.1038/ncpgasthep0259. PMID 16265432
- [Result] Biyikoglu I, Babali A, Cakal B, Koklu S, Filik L, Astarci MH, Ustun H, Ustundag Y, Akbal E. Do scattered white spots in the duodenum mark a specific gastrointestinal pathology? J Dig Dis. 2009 Nov;10(4):300-4. doi: 10.1111/j.1751-2980.2009.00399.x. PMID 19906109